CLINICAL TRIAL: NCT05413057
Title: A Multicenter, Prospective, Observational Study to Evaluate Effectiveness and Safety of Fixed-dose Combinations of Fimasartan/Amlodipine or Fimasartan/Amlodipine/Hydrochlorothiazide in Essential Hypertensive Patients
Brief Title: An OS to Evaluate Effectiveness and Safety of Fixed-dose Combinations of FMS/AML or FMS/AML/HCTZ
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-408
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension,Essential
Keywords: Fimasartan; Essentail hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this observation study is to collect data on the effects and side effects for 12 weeks of the medication administration of the single-pill combinations, which are fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide, based on fimasartan. (Stage 1).

Also, this study will evaluate major cardiovascular events, long-term blood pressure control, and the safety by follow-up of those who consent to the extended study for about 2 years (96 weeks).(Stage 2)

DETAILED DESCRIPTION:
This study will be conducted as a prospective observational study in about 600 domestic medical institutions, which are at least clinical level.

The investigator will enroll those who have essential hypertension and meet the inclusion and exclusion criteria after obtaining voluntary written consent for participation in the study and use of personal information.

This study is a non-interventional observational study and is based on decisions by the investigator about the choice of antihypertensive drugs, the period of treatment, and the medication change status etc.

During this study period, the scope of data to be collected is as follows:

* Demographic information
* Disease information (historical diseases and concomitant diseases )
* Physical measurements and vital signs
* Blood pressure Central Blood pressure and hemodynamic values (if applicable)
* Information on antihypertensive drugs and other concomitant medications
* Adverse drug reaction(ADR) and serious adverse drug reactions(SADR) related to fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide
* Information on cardiovascular events (Only if subjects are in long term follow-up)
* Death information (Only if subjects are in long term follow-up)

ELIGIBILITY:
* Inclusion Criteria:

  1. Patients who voluntarily consent on the informed consent form and understand the study's purpose, methods, and so on
  2. Males and females over the age of 19
  3. Patients who have been diagnosed with essential hypertension and plan to be treated with fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide

     If the patient is applicable, one of the following;
     * If the patients have severe hypertension, stage 2 or higher(sit SBP ≥ 160 mmHg or sit DBP ≥ 100 mmHg), or high-risk hypertension (The cardiovascular risk score of the 2018 hypertension treatment guidelines by the Korean Society of Hypertension is applied.) The patients have never been treated with antihypertensive drugs for essential hypertension.
     * If the patients are on concomitant administration of fimasartan/amlodipin and hydrochlorothiazide for essential hypertension or, If the patients are on concomitant administration of a fimasartan/hydrochlorothiazide combination and amlodipine for essential hypertension
     * If the patients have a blood pressure of sitSBP ≥ 140 mmHg or sitDBP ≥ 90 mmHg even though they have been treated with antihypertensive drugs for essential hypertension
  4. The patients who understand this study and are available to participate in this study until the end of the study period with a cooperative attitude.
* Exclusion Criteria:

  1. The patients who are suspected of having secondary hypertension or confirmed to have secondary hypertension
  2. The patients who are contraindicated to taking fimasartan complex according to the drug labelling
  3. The patients who are currently participation in another clinical trials (Drugs or medical devices) The patients who took an investigational drug within 12 weeks of the enrollment date

     However, the following patients can participate in this study:

     The patients who are currently enrolled in non-interventional clinical studies or who are being followed up on after the administration of investigational drugs has ended.
  4. The patients who are not suitable for this study by the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Essential hypertensive patients in need of a combination treatment with two or more antihypertensive agents
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The blood pressure control rate | Week 12
  The blood pressure control rate (< 140/90 mmHg)(Systolic and Diastolic) at Week 12

SECONDARY OUTCOMES:
The blood pressure control rate | Week 8
  The blood pressure control rate (< 140/90 mmHg) at Week 8
The target blood pressure control rate | Week 12
  The target blood pressure control rate (< 140/90 mmHg) at Week 12
Change in central systolic pressure(CSP) and Central diastolic pressure(CDP) | Week 12
  Change in central systolic pressure(CSP) and Central diastolic pressure(CDP) at Week 12 from baseline (Only the subjects who measured the central blood pressure)
Control rate of The Blood pressure control rate | Week 36, Week 48, Week 96
  Control rate of The Blood pressure control rate(< 140/90 mmHg) at Week 36 , 48 and 96
The target blood pressure control rate | Week 36, Week 48, Week 96
  The target blood pressure control rate at Week 36 , 48 and 96
The incidence rate of major cardiovascular event(MACE) | Week 96
  The incidence rate of major cardiovascular event(MACE)

OTHER OUTCOMES:
Adverse drug reactions(ADR) related to fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide | Week 12, Week 96
  Adverse drug reactions(ADR) related to fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide (From the baseline to Week 12, From the baseline to Week 96)
Serious Adeverse Drug Reaction(Serious ADR) related to fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide | Week 12, Week 96
  Serious Adeverse Drug Reaction(Serious ADR) related to fimasartan/amlodipine or fimasartan/amlodipine/hydrochlorothiazide (From the baseline to Week 12, From the baseline to Week 96)

CONTACTS AND LOCATIONS:
Overall Officials: MyungSook Hong, Study Director — Boryung Co.,Ltd.
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No